CLINICAL TRIAL: NCT04988009
Title: Patient Perceptions Around Quality of Care Through Telemedicine in Neuro-Oncology
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0493; NCI-2020-07493 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0493 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-07; First posted 2021-08-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Central Nervous System Neoplasm; Leptomeningeal Neoplasm; Metastatic Malignant Neoplasm in the Brain; Primary Brain Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningeal Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey, medical chart review): Patients complete a survey related to their perceived quality of care via telephone and have their medical chart reviewed prospectively.
  Interventions: Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical chart
Other: Survey Administration — Complete survey

SUMMARY:
This study evaluates patient perceptions around quality of care through telemedicine in neuro-oncology. Studying questionnaires related to perceptions quality of care through telemedicine in patients with brain cancer may help doctors to improve the delivery of care through this modality.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the patient-perceived quality of care by group (telemedicine versus in-person visits) in patients with central nervous system (CNS) cancer.

SECONDARY OBJECTIVES:

I. To characterize the visits provided by telemedicine compared to those in-person.

II. To contrast the average time spent on telemedicine visits compared to in-person visits, and the delay between visit order placement and visit occurring.

III. To evaluate the domains of patient care addressed on a telemedicine visit versus in-person visit per documentation, including (1) treatment planning, (2) symptom burden, (3) goals of care.

IV. To evaluate frequency of acute care sought (through emergency room or urgent care clinic) within 30 days of encounter in telemedicine visit versus (vs) in-person visit.

V. The impact of patient and clinical characteristics on perceived quality of care in the context of covariate-adjusted modeling.

OUTLINE:

Patients complete a survey related to their perceived quality of care via telephone and have their medical chart reviewed prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a CNS tumors: this includes patients with primary brain tumors, brain metastases, and leptomeningeal disease
* Established patients with a follow up encounter with Neuro-Oncology at the Brain and Spine Center at the University of Texas MD Anderson Cancer Center; this encounter can be

  * An in-person visit
  * A telemedicine appointment

Exclusion Criteria:

* Encounter occurred with the assistance of official language translation support
* Patients with telephone encounters (without interactive video)
* New patient or consult visits
* Neither patient nor caregiver present during the visit are available or able to answer survey questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with encounters at the Brain and Spine Center between 4/20/2020 and either (1) 8/30/2020 or (2) date that the state of emergency secondary to the COVID-19 pandemic is declared terminated in the United States of America- whichever date is earlier
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survey response to question 6 of the quality of care survey ("I felt I received good medical care during this encounter") | through study completion, an average of 1 year
  Survey responses will be summarized by ordinal category as counts with percentages, separately by group. Will separately estimate the proportion of each ordinal level of each group with 95% confidence interval.

SECONDARY OUTCOMES:
Quality of Care Survey | through study completion, an average of 1 year
  Will separately estimate the proportion of each ordinal level of each group with 95% confidence interval.
Patients and clinical characteristics | Baseline
  Differences between groups will be assessed by 2-sample 2-sided t-test and Mann-Whitney test, Fisher's exact test, or chi-square test.
Interactive time spent during visit | through study completion, an average of 1 year
  Will be summarized by group per mean, median, standard deviation, and range. Differences between groups will be assessed by t-test and Mann-Whitney test.
Time from visit order placement to visit occurring | through study completion, an average of 1 year
  Will be summarized by group per mean, median, standard deviation, and range. Differences between groups will be assessed by t-test and Mann-Whitney test.
Domains of patient care addressed during a visit, including treatment planning, symptom burden, and goals of care | through study completion, an average of 1 year
  Will be summarized as counts with percentages by group. Differences between groups will be assessed by chi-square test.
Incidence of acute care sought (through emergency room or urgent care clinic) | Within 30 days of encounter
  Will be summarized as counts with percentages by group. Differences between groups will be provisionally assessed by Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J O'Brien, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org